CLINICAL TRIAL: NCT06678607
Title: Phase I Clinical Trial to Evaluate the Safety and Tolerability of 24-valent Pneumococcal Polysaccharide Conjugate Vaccine in People Aged 18 Years and Older
Brief Title: Phase I Clinical Trial of PCV24 in People Aged 18 Years and Older
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Reinovax Biologics Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: JSVCT182
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Pneumococcal Infectious Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental group 1 (Experimental): 60 participants will be randomized to receive Reinovax PCV24 formulation 1. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Reinovax PCV24 formulation 1
- Experimental group 2 (Experimental): 60 participants will be randomized to receive Reinovax PCV24 formulation 2. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Reinovax PCV24 formulation 2
- Active control group (Active Comparator): 60 participants will be randomized to receive PPSV23. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: PPSV23
- Placebo group (Placebo Comparator): 60 participants will be randomized to receive placebo. The route of administration is intramuscular injection at the deltoid muscle of the upper arm. The immunization schedule is 1 dose.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Reinovax PCV24 formulation 1 — One dose of Reinovax PCV24 formulation 1（0.5mL）
  Arms: Experimental group 1
Biological: Reinovax PCV24 formulation 2 — One dose of Reinovax PCV24 formulation 1（0.5mL）
  Arms: Experimental group 2
Biological: PPSV23 — One dose of PPSV23 (0.5 mL) contains 1、2、3、4、5、6B、7F、8、9N、9V、10A、11A、12F、14、15B、17F、18C、19A、19F、20、22F、23F and33F saccharides.
  Arms: Active control group
Biological: Placebo — One dose of 0.5 mL placebo is aluminum phosphate adjuvant (aluminum content 0.25mg/dose), sodium chloride, succinic acid, polysorbate 80, and water for injection except for antigen components in 24-valent pneumococcal polysaccharide conjugate vaccine
  Arms: Placebo group

SUMMARY:
Phase I clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Shanghai Reinovax Biologics Co., LTD will be conducted in Chinese adults aged 18 years and older . The objective of the study is to evaluate the safety and tolerability of PCV24. The trial is a single-center, randomized, blind,parallel-controlled design I clinical trial.

DETAILED DESCRIPTION:
Phase I clinical trial of 24-valent pneumococcal conjugate vaccine (PCV24) developed by Shanghai Reinovax Biologics Co., LTD will be conducted in Chinese adults aged 18 years and older. The objective of the study is to evaluate the safety and tolerability of PCV24. The active control vaccine is a 23-valent pneumococcal polysaccharide vaccine (23-valent pneumococcal polysaccharide vaccine, PPSV23) produced by the Chengdu Institute of Biological Products. The placebo is aluminum phosphate adjuvant (aluminum content 0.25mg/dose), sodium chloride, succinic acid, polysorbate 80, and water for injection except for antigen components in 24-valent pneumococcal polysaccharide conjugate vaccine developed by Shanghai Ruizhou Biotechnology Co., Ltd. and Vinorelite Biopharmaceutical Co., Ltd.

A total of at least 240 participants will be enrolled, including 84 adults aged 18-60years and 120 elderly people aged ≥61 years. Participants will be randomized in a 1:1:1:1 ratio to receive one dose of PCV24 formulation 1, PCV24 formulation 2, PPSV23 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers over the age of 18 on the day of screening, and can provide legal identification;
2. Informed consent must be obtained from the volunteer and signed informed consent form;
3. Volunteers are able and willing to comply with the requirements of the clinical trial protocol and can attend all visits;
4. Armpit body temperature ≤ 37.0 °C on the day of enrollment.

Exclusion Criteria:

1. Previous pneumococcal vaccination, or history of invasive disease caused by pneumococcal in the past;
2. Have any previous history of severe allergies to vaccines or drugs, such as anaphylactic shock, allergic laryngeal edema, Henoch-Schonlein purpura, thrombocytopenic purpura, local allergic necrosis reaction (Athus reaction), etc.;
3. Have been diagnosed with congenital or acquired immunodeficiency, or have recently received immunosuppressant therapy, such as systemic glucocorticoid therapy such as prednisone or similar drugs > 5 mg/day for more than 2 consecutive weeks in 1 month before vaccination (Note: the use of topical and inhaled/nebulized steroids can participate);
4. Suffering from serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension that cannot be controlled by medication (when measured on site: systolic blood pressure ≥ 160 mmHg, diastolic blood pressure ≥100 mmHg), etc.;
5. Suffering from acute febrile illness or infectious diseases, such as tuberculosis, viral hepatitis, etc.;
6. History of nervous system damage, severe congenital malformations, severe developmental disabilities, severe genetic defects, severe malnutrition, etc.;
7. Have a history or family history of epilepsy, encephalopathy, or psychiatric disorders;
8. Those who have been diagnosed with thrombocytopenia, any abnormal coagulation function (such as coagulation factor deficiency, coagulation disorders, platelet abnormalities, etc.) or contraindications to intramuscular injection such as anticoagulant therapy;
9. asplenia, functional asplenia, and asplenia or splenectomy due to any cause;
10. Suffering from severe chronic diseases or conditions that cannot be controlled smoothly in the advanced stage, such as diabetes, thyroid disease, etc.;
11. Have received blood or blood-related products or immunoglobulins within 3 months;
12. Received live attenuated vaccine within 14 days;
13. Received other vaccines within 7 days;
14. Received other investigational drugs or vaccines within 1 month;
15. Is participating in or plans to participate in clinical studies of other drugs or vaccines during the study period;
16. Any other condition that, in the opinion of the investigator, may interfere with the study evaluation;
17. Those who have abnormal laboratory tests such as blood routine, blood biochemistry, and urine routine that are clinically significant and cannot be enrolled according to the comprehensive judgment of the investigator;
18. Exclusion Criteria for Partial Populations:

Females of childbearing potential (18~49 years old): positive urine pregnancy test on the day of enrollment, lactation, or pregnancy plans within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2023-11-19 (Actual); Primary Completion 2024-07-28 (Actual); Study Completion 2024-07-28 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse reactions | 0-7days after vaccination
  Incidence of adverse reactions within 7 days after vaccination

SECONDARY OUTCOMES:
incidence of adverse events | 0~30 days after vaccination.
  The incidence of adverse events within 30 days after vaccination.
Incidence of serious adverse events (SAE) | 0-6 months after vaccination
  Incidence of SAE during the period of safety monitoring
Incidence of clinically significant abnormality in laboratory examination tests | 0-3days after vaccination
  Incidence of clinically significant abnormality in blood routine, blood biochemistry,coagulation function and urine routine test results within 3 days after vaccination

CONTACTS AND LOCATIONS:
Locations (1):
- Zhenjiang Center for Disease Control and Prevention, Zhenjiang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No